CLINICAL TRIAL: NCT04368923
Title: Management of Covid-19 Patients During Home Isolation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Sedky, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/012-2020
Record Dates: First submitted 2020-04-24; First posted 2020-04-30 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Covid 19
MeSH Terms: conditions — COVID-19 | interventions — Oxygen Inhalation Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxygen Therapy Group (Experimental)
  Interventions: Device: Oxygen Therapy
- Physical Therapy Group (Experimental)
  Interventions: Procedure: Physical Therapy

INTERVENTIONS:
Device: Oxygen Therapy — Patients receive oxygen therapy
  Arms: Oxygen Therapy Group
Procedure: Physical Therapy — Patients receive physical therapy
  Arms: Physical Therapy Group

SUMMARY:
This study will be concerned with managing patients of Covid-19 while being home isolated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Covid-19
* American Society of Anesthesiologists (ASA) class I
* >= 21 years old
* <= 40 years old

Exclusion Criteria:

* ASA class II, class III or class IV

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-06-21 (Estimated); Study Completion 2020-06-23 (Estimated)

PRIMARY OUTCOMES:
Arterial Blood Gases (ABG): Partial Pressure of Oxygen and Carbon Dioxide | 48 hours
Arterial Blood Gases (ABG): Acidity Potential Hydrogen (pH) | 48 hours

SECONDARY OUTCOMES:
Vital Signs (Temprature) | 24 hours
Vital Signs (Respiratory Rate) | 24 hours
Vital Signs (Oxygen Saturation) | 24 hours
Vital Signs (Heart Rate) | 24 hours
Vital Signs (Blood Pressure) | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- M. Sedky, Cairo, Egypt

REFERENCES:
- [Derived] Adly AS, Adly MS, Adly AS. Telemanagement of Home-Isolated COVID-19 Patients Using Oxygen Therapy With Noninvasive Positive Pressure Ventilation and Physical Therapy Techniques: Randomized Clinical Trial. J Med Internet Res. 2021 Apr 28;23(4):e23446. doi: 10.2196/23446. PMID 33819166